CLINICAL TRIAL: NCT05139550
Title: Smartphone Rehabilitation App For Stroke Survivor
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Riphah International University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: REC/00828 Rabiya Tahir
Record Dates: First submitted 2021-10-26; First posted 2021-12-01 (Actual); Last update posted 2022-04-18 (Actual); Status verified 2022-04

CONDITIONS: Stroke
Keywords: stroke; CVA
MeSH Terms: conditions — Stroke

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Smartphone Rehabilitation Application (Experimental): Upper Limb Exercise Protocol:
  Passive Exercises ROMs for shoulder, ROMs for elbow, ROMs for wrist,fingers and thumb
  Active/Assisted Exercises bilateral shoulder flexion with both hands interlocked, Elbow pronation and supination, Wrist flexion and extension with the help of unaffected hand, Forearm to box, Extend elbow (side), Hand to box (front)
  Functional Activities Lift can, Lift pencil, Lift paper clip, Stack checkers, Flip cards, Fold towel, drinking water from a glass, lifting a glass of water to a level of 90° shoulder flexion with an extended elbow, moving 5 crystals from the table to a box, wiping the table with a towel with the elbow extended, grasping and releasing a 6 cm in diameter tennis ball, combing their hair, Eating with affected hand, opening and closing jars
  Interventions: Device: Smartphone Rehabilitation Application

INTERVENTIONS:
Device: Smartphone Rehabilitation Application — Upper Limb Exercise Protocol:
  Passive Exercises
  ROMs for shoulder, ROMs for elbow, ROMs for wrist,fingers and thumb
  Active/Assisted Exercises
  bilateral shoulder flexion with both hands interlocked, Elbow pronation and supination, Wrist flexion and extension with the help of unaffected hand, Forearm to box, Extend elbow (side), Hand to box (front)
  Functional Activities
  Lift can, Lift pencil, Lift paper clip, Stack checkers,Flip cards, Fold towel, drinking water from a glass, lifting a glass of water to a level of 90° shoulder flexion with an extended elbow, moving 5 crystals from the table to a box, wiping the table with a towel with the elbow extended, grasping and releasing a 6 cm in diameter tennis ball, combing their hair, Eating with affected hand, opening and closing jars

SUMMARY:
This is a pilot study of a smartphone app in which the tool will be developed and validation of the tool will be done for the rehabilitation of upper limb in stroke survivors. The study will be divided into two phases. The first phase will be the development of a smartphone app for upper limb function. The second phase of the study will be a pilot study where 10 stroke patients will be recruited and upper limb intervention will be applied through a smartphone app.

ELIGIBILITY:
Inclusion Criteria:

* Subacute and chronic stroke patient > 3 months post stroke till 1 year.
* Modified Ashworth scale scoring ≤ 2
* An ability to understand the command
* First ever stroke
* Grade II, III on Functional mobility Scale
* Able to use and comprehend smart phone.

Exclusion Criteria:

* Vestibular disorders, paroxysmal vertigo
* Presence of other neurological conditions such as neglect, hemianopsia and pushing syndrome

Ages: 40 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2021-11-21 (Actual); Primary Completion 2022-01-30 (Actual); Study Completion 2022-02-22 (Actual)

PRIMARY OUTCOMES:
Wolf Motor Function Test (WMFT) | 4 weeks
  The Wolf Motor Function Test (WMFT) quantifies upper limb motor ability through timed and functional tasks. Original WMFT contains 21 items but widely used WMFT contains 17 items.
  The maximum time allowed for each task is 120 seconds. Each task is rated on a 6 point scale of 0-5 0 means unable to attempt the task while 5 means normal. Lower scores indicate lower functioning levels.
Nine-Hole Peg Test (9HPT) | 4 weeks
  The Nine-Hole Peg Test (9HPT) is used to measure finger dexterity in various neurological conditions.
  Patients are scored in seconds based on the time taken to complete the activity. The stopwatch should be started from the moment the participant touches the first peg until the moment the last peg hits the container.
  Alternative scoring - the number of pegs placed in 50 or 100 seconds can be recorded. In this case, results are expressed as the number of pegs placed per second

CONTACTS AND LOCATIONS:
Overall Officials: Aruba Saeed, PhD*, Study Chair — Riphah International University
Locations (1):
- Riphah International University, Rawalpindi, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: No